CLINICAL TRIAL: NCT01391325
Title: Long-term Allopurinol Safety Study Evaluating Outcomes in Gout Patients (LASSO)
Brief Title: Allopurinol Outcome Study
Acronym: LASSO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-401
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allopurinol (Other): Treatment.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Allopurinol — Commercially available allopurinol 100 mg and 300 mg oral tablets will be prescribed by the Investigator according to the approved product label.

SUMMARY:
This is a study of allopurinol in gout patients with hyperuricemia that will evaluate the safety and serum urate (sUA) lowering capability of allopurinol as a urate lowering therapy (ULT) for up to six months. Allopurinol will be dosed according to the local product label, at the discretion of the Investigator, to achieve an optimal, medically appropriate dose for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnosis of gout according to the American Rheumatism Association (ARA) Criteria for the Classification of Acute Arthritis of Primary Gout.
* Not on a urate lowering therapy (ULT) must have an sUA level ≥ 8.0 mg/dL at screening.
* If on concomitant ULT must have an sUA level ≥ 6.5 mg/dL at screening.
* Must have had at least 2 gout flares in the past year.

Exclusion Criteria:

* Consumption of more than 14 drinks of alcohol per week (eg, 1 drink = 5 oz [150 mL] of wine, 12 oz [360 mL] of beer, or 1.5 oz [45 mL] of hard liquor).
* History or suspicion of drug abuse.
* History of autoimmune disease requiring systemic treatment.
* Known or suspected human immunodeficiency virus (HIV), hepatitis C antibody (HCV), or hepatitis B antibody (HBsAg) infection.
* History of malignancy within the previous 5 years (with the exception of nonmelanoma skin cancer that has been treated with no evidence of recurrence, treated cervical dysplasia or treated in situ Grade 1 cervical cancer).
* Myocardial infarction, unstable angina, New York Heart Association (NYHA) class III or IV heart failure, or stroke within the last 12 months.
* Uncontrolled hypertension (systolic pressure above 160 mm Hg or diastolic pressure above 95 mm Hg).
* Estimated creatinine clearance < 30 mL/min by Cockcroft-Gault formula.
* Kidney or other organ transplant.
* Active peptic ulcer disease requiring treatment.
* History of xanthinuria, active liver disease, or hepatic dysfunction.
* If unable to take gout flare prophylaxis of either colchicine or nonsteroidal anti-inflammatory drugs (NSAIDs) due to contraindication (e.g. toxicity, renal function, use of contraindicated medications).
* Known hypersensitivity or allergy to allopurinol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1735 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S Baumgartner, MD, Study Director — Ardea Biosciences, Inc.
Locations (158):
- United States (116):
  - Birmingham, Alabama
  - Bringham, Alabama
  - Calera, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Chandlers, Arizona
  - Green Valley, Arizona
  - Jonesboro, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Carmichael, California
  - Covina, California
  - Hemet, California
  - Irvine, California
  - Los Angeles, California
  - Mission Viejo, California
  - Pasadena, California
  - Sacramento, California
  - San Diego, California
  - San Ramon, California
  - Santa Maria, California
  - Weslake Village, California
  - Denver, Colorado
  - Englewood, Colorado
  - Danbury, Connecticut
  - Trumbull, Connecticut
  - Brandenton, Florida
  - Brandon, Florida
  - Brooksville, Florida
  - East Brandenton, Florida
  - Fleming Island, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Oldsmar, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Plant City, Florida
  - Port Orange, Florida
  - Sanford, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Winter Haven, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Newnan, Georgia
  - Honolulu, Hawaii
  - Meridian, Idaho
  - Addison, Illinois
  - Chicago, Illinois
  - Gurnee, Illinois
  - Evansville, Indiana
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Monroe, Louisiana
  - Cumberland, Maryland
  - Frederick, Maryland
  - Hagerstown, Maryland
  - Wheaton, Maryland
  - Hyannis, Massachusetts
  - Worcester, Massachusetts
  - South Traverse City, Michigan
  - Rochester, Minnesota
  - Olive Branch, Mississippi
  - Florissant, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Nashua, New Hampshire
  - Albuquerque, New Mexico
  - Albany, New York
  - Endwell, New York
  - Hartsdale, New York
  - Charlotte, North Carolina
  - Harrisburg, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Altoona, Pennsylvania
  - Duncansville, Pennsylvania
  - Lancaster, Pennsylvania
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Spartanburg, South Carolina
  - Jackson, Tennessee
  - Spring Hill, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Irving, Texas
  - Mesquite, Texas
  - San Antonio, Texas
  - Sugar Land, Texas
  - Bountiful, Utah
  - West Jordan, Utah
  - Arlington, Virginia
  - Richmond, Virginia
  - Port Orchard, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Morgantown, West Virginia
- Australia (11):
  - Camperdown, New South Wales
  - Wollongong, New South Wales
  - Birsbane, Queensland
  - Daw Park, South Australia
  - Woodville South, South Australia
  - Hobart, Tasmania
  - Clayton, Victoria
  - Heidelberg, Victoria
  - North Ballarat, Victoria
  - Perth, Western Australia
  - Malvern East
- Belgium (5):
  - Brussels
  - Gozée
  - Kortrijk
  - Mouscron
  - Yvoir
- Canada (7):
  - Coquitlam, British Columbia
  - Kelowna, British Columbia
  - Penticton, British Columbia
  - Ottawa, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Québec, Quebec
- Germany (3):
  - Altenburg
  - Dresden
  - Eichstätt
- New Zealand (6):
  - Christchurch, Canterbury
  - Auckland
  - Hamilton
  - Papatoetoe
  - Rotorua
  - Tauranga
- South Africa (10):
  - Bloemfontein
  - Durban
  - East London
  - Johannesburg
  - Paarl
  - Pretoria
  - Rondebosch
  - Stellenbosch
  - Thabazimbi
  - Worcester

REFERENCES:
- [Derived] Topless R, Noorbaloochi S, Merriman TR, Singh JA. Change in serum urate level with urate-lowering therapy initiation associates in the immediate term with patient-reported outcomes in people with gout. Semin Arthritis Rheum. 2022 Oct;56:152057. doi: 10.1016/j.semarthrit.2022.152057. Epub 2022 Jun 29. PMID 35835008
- [Derived] Becker MA, Fitz-Patrick D, Choi HK, Dalbeth N, Storgard C, Cravets M, Baumgartner S. An open-label, 6-month study of allopurinol safety in gout: The LASSO study. Semin Arthritis Rheum. 2015 Oct;45(2):174-83. doi: 10.1016/j.semarthrit.2015.05.005. Epub 2015 May 21. PMID 26190562

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1,735 subjects enrolled in the study; however, only 1,732 were treated. Therefore, 1,732 subjects started the treatment period.
Period: Overall Study
Arm/Group | Allopurinol
Started | 1732
Completed | 1238
Not Completed | 494

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of allopurinol.
Arm/Group | Allopurinol
Number analyzed (Participants) | 1732
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years at enrollment.
  years | 51.4 (11.93)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1483
  >=65 years | 249
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 1614
Region of Enrollment [Number; unit: participants]
  United States | 1203
  Canada | 74
  Belgium | 11
  Australia | 104
  South Africa | 242
  Germany | 14
  New Zealand | 84

OUTCOME MEASURES:

1. Primary Outcome: Safety of Allopurinol
Description: Proportion of subjects who experienced at least one Treatment Emergent Adverse Event (TEAE) during the study.
Time Frame: Every month for 6 months.
Population: All subjects who received at least one dose of allopurinol
Measure: Number; unit: percentage of subjects
Arm/Group | Allopurinol
Number analyzed (Participants) | 1732
percentage of subjects | 55.1

2. Secondary Outcome: Proportion of Subjects With Serum Urate (sUA) Less Than 6.0 mg/dL
Description: Proportion of subjects with serum urate (sUA) less than 6.0 mg/dL at Month 6 using Last Observation Carried Forward (LOCF) for subjects with missing values at Month 6.
Time Frame: Month 6
Population: All subjects who received at least one dose of allopurinol
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Allopurinol
Number analyzed (Participants) | 1732
percentage of subjects | 43.4 [41.0 to 46.0]

3. Secondary Outcome: Incidence of Gout Flares
Description: Proportion of subjects who experienced at least one gout flare requiring treatment during the study.
Time Frame: Every month for 6 months.
Population: Subjects who received at least one dose of allopurinol
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Allopurinol
Number analyzed (Participants) | 1732
percentage of subjects | 33.4 [31.0 to 36.0]

4. Secondary Outcome: Mean Change From Baseline to Month 6 in SF-36 PCS+MCS
Description: The SF-36 is a short-form health survey with 36 questions that yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical (PCS) and mental health (MCS) summary. Each scale is directly transformed into a 0-100 scale. The lower the score the more disability. The higher the score the less disability. The component scores (PCS and MCS) are norm-based to a standard population with a mean of 50 and a standard deviation of 10.
Time Frame: Month 6
Population: Subjects who recieved at least one dose of allopurinol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Allopurinol
Number analyzed (Participants) | 1732
units on a scale
  SF-36 Physical Component Summary | 3.88 (8.458)
  SF-36 Mental Health Component Summary | 0.71 (9.076)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Allopurinol
Serious Adverse Events (participants affected / at risk) | 52/1732
Other Adverse Events (participants affected / at risk) | 654/1732
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allopurinol (N=1732)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pericarditis constrictive (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Death (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Abscess intestinal (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Cholecystitis infective (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Perirectal abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Pancreatic enzymes increased (Investigations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 2 (2)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 1 (1)
Breathing-related sleep disorder (Psychiatric disorders) | 1 (1)
Panic disorder with agoraphobia (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Allopurinol (N=1732)
Upper Respiratory Tract Infection (Infections and infestations) | 100
Diarrhoea (Gastrointestinal disorders) | 77
Athralgia (Musculoskeletal and connective tissue disorders) | 55
Nasalphrayngitis (Infections and infestations) | 53
Blood creatine phosphokinase increased (Investigations) | 48
Back pain (Musculoskeletal and connective tissue disorders) | 45
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44
Hypertension (Vascular disorders) | 43
Headache (Nervous system disorders) | 41
Alanine aminotransferase increased (Investigations) | 38
Bronchitis (Infections and infestations) | 29
Influenza (Infections and infestations) | 26
Rash (Skin and subcutaneous tissue disorders) | 26
Muscle strain (Injury, poisoning and procedural complications) | 25
Nausea (Gastrointestinal disorders) | 24
Aspartate aminotransferase increased (Investigations) | 23
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20
Urinary tract infection (Infections and infestations) | 19
Liver function test abnormal (Investigations) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.